CLINICAL TRIAL: NCT06241846
Title: A Multicenter, Open-Label, Phase II Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of YL201 in Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Phase II Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of YL201 in Patients With mCRPC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MediLink Therapeutics (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YL201-CN-201-01
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Castration-resistant Prostate Cancer (mCRPC)
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1 (Experimental): To evaluate the safety and efficacy of YL201 in patients with mCRPC and to determine the recommended dose of YL201 for the pivotal clinical study (n ≈ 60)； Cohort 1: YL201 2.0 mg/kg iv Q3W ； Cohort 2: YL201 1.6 mg/kg iv Q3W； Cohort 3: YL201 2.4 mg/kg iv Q3W； Cohort 4: YL201 1.2 mg/kg iv D1, D8 Q3W； Cohort 5: YL201 1.0 mg/kg iv D1, D8, Q3W；
  Interventions: Drug: YL201 for Injection
- Part2 (Experimental): To evaluate the safety and efficacy of YL201 in patients with mCRPC and to determine the recommended dose of YL201 for the pivotal clinical study (n ≈ 40)； Recommended dose and method of administration
  Interventions: Drug: YL201 for Injection

INTERVENTIONS:
Drug: YL201 for Injection — Patients will be treated with YL201 intravenous (IV) infusion once every 3 weeks on Day 1 or twice every 3 weeks on Day 1 and Day 8 during a 3-week (21-day) cycle.

SUMMARY:
This is a multicenter, open-label, phase II study of YL201 in China to evaluate the efficacy, safety, and PK characteristics of YL201 on mCRPC.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who understand relevant information of the study prior to initiation of the study and voluntarily sign and date on the ICF.
2. Age ≥ 18 years.
3. Patients should meet the following conditions to be enrolled:

   * Histologically or cytologically confirmed prostate cancer. Note: The primary histological classification indicated by biopsy should be adenocarcinoma;
   * Meeting the following criteria for clinical diagnosis of mCRPC:

<!-- -->

1. Subjects who understand relevant information of the study prior to initiation of the study and voluntarily sign and date on the ICF.
2. Age ≥ 18 years.
3. Patients should meet the following conditions to be enrolled:

   • Histologically or cytologically confirmed prostate cancer. Note: The primary histological classification indicated by biopsy should be adenocarcinoma;

   • Meeting the following criteria for clinical diagnosis of mCRPC:

   √Testosterone level after castration (a serum testosterone level of <50 ng/dl or 1.7 nmol/L);
   * Serum prostate specific antigen (PSA) progression (PSA > 1 ng/mL and 2 consecutive increases in PSA with at least a 1-week interval >50% from baseline), or PD by imaging (≥ 2 new bone lesions suggested by a bone scan according to PCWG3 criteria; and/or progression of soft tissue lesions suggested by computed tomography (CT) or nuclear magnetic resonance imaging (MRI) according to RECIST v1.1); meeting either or both criteria;
   * Persistent luteinizing hormone-releasing hormone (LHRH) analogue castration (medical castration) or prior bilateral orchiectomy (surgical castration); surgical castration should be performed at least 3 months prior to enrollment, and medical castration is required from at least 3 months prior to the first dose and throughout the study for subjects not yet undertake bilateral orchiectomy; • Patients with progression on or intolerance to at least one prior novel hormone therapy (NHT) (e.g., enzalutamide, abiraterone, darolutamide, apalutamide, or rezvilutamide); • Prior therapy with no more than 2 lines of chemotherapy is allowed; • Patients with known previous prostate adenocarcinoma with a documented BRCA1/2 (germline or somatic) mutation should have received poly ADP ribose polymerase (PARP) inhibitor therapy (if available and tolerated);
4. Patients with metastatic lesions confirmed by CT, MRI, or bone scan imaging within 28 days prior to the first dose.
5. Patients with archived or fresh tumor tissue samples. Patients who cannot provide tumor samples or cannot provide sufficient samples may be enrolled in this study after considering specific circumstances and discussions with the Sponsor.

   • Fresh tumor tissue samples (formalin-fixed, paraffin-embedded (FFPE) tumor blocks or FFPE sections) should be provided for retrospective detection of B7H3 expression by the central laboratory using the immunohistochemistry [IHC] method; if fresh tumor tissue samples are not available, FFPE tumor blocks previously archived are acceptable, and fresh FFPE sections should be prepared within 2 weeks.
6. Eastern cooperative oncology group performance status (ECOG PS) score of 0 or 1.
7. The function of organs and bone marrow meets the requirements within 7 days prior to the first dose, which is defined as follows:

   • Hemoglobin (Hb) ≥ 90 g/L (no blood transfusion or erythropoietin treatment within 14 days prior to the first dose);

   • Absolute neutrophil count (ANC) ≥ 1.5×109/L (no treatment with granulocyte colony stimulating factor or granulocyte-macrophage colony stimulating factor within 14 days prior to the first dose);

   • Platelet count (PLT) ≥ 100×109/L (no platelet transfusion, thrombopoietin, or interleukin-11 within 14 days prior to the first dose);

   • Total bilirubin (TBIL) ≤ 1.5×upper limit of normal (ULN) in the absence of obvious liver metastasis, or ≤ 3×ULN in the presence of liver metastasis;

   • Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3×ULN in the absence of obvious liver metastasis or ≤ 5×ULN in the presence of liver metastasis;

   • Serum albumin (ALB) ≥ 30 g/L;

   • Creatinine clearance calculated using Cockcroft-Gault formula ≥ 50 mL/min or the creatinine ≤ 1.5×ULN;
   * Activated partial thromboplastin time (APTT) and international normalized ratio (INR) ≤ 1.5×ULN, except for patients who are on anticoagulant therapy. In this case, a stable anticoagulant regimen should be maintained with APTT and INR controlled within the range deemed appropriate by the investigator.
8. Patients must agree to adopt highly effective contraceptive measures from screening, throughout the study period, and within at least 6 months after the last dose of the investigational drug.
9. Expected survival ≥ 6 months.
10. Be capable of and willing to comply with the visits and procedures stipulated in the study protocol.

Exclusion Criteria:

1. Previously treated with drugs targeting B7H3.
2. Currently participating in another clinical study, unless it is an observational (non-interventional) clinical study, or the patient is at the follow-up period of an interventional study.
3. Previously treated with topoisomerase I inhibitors or ADC therapy composed of topoisomerase I inhibitors.
4. The washout period of the previous anti-tumor therapy is considered insufficient.
5. Patients received major surgery.
6. Prior treatment with allogeneic bone marrow transplantation or solid organ transplantation.
7. Prior treatment with glucocorticoids for more than 28 consecutive days within 28 days prior to the first dose of the investigational drug.
8. Patients received any live vaccine within 4 weeks prior to the first dose of the investigational drug, or plan to receive live vaccine during the study period.
9. Have pathological long bone fracture, or the risk of pathological long bone fracture.
10. Have meningeal metastasis or cancerous meningitis.
11. Have uncontrolled bladder outlet obstruction or urinary incontinence.
12. Have brain metastasis or spinal cord compression.
13. Patients with uncontrolled or clinically significant cardiovascular diseases.
14. Clinically significant complicated pulmonary disorders.
15. Diagnosed with Gilbert's syndrome.
16. Accompanying uncontrolled effusion in the third space requiring repeated drainage.
17. Medical history of gastrointestinal perforation and/or fistula within 6 months prior to the first dose, or active gastric and duodenal ulcers, ulcerative colitis, or other gastrointestinal diseases that may cause hemorrhage or perforation in the opinion of the investigator.
18. Active serious infection (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] ≥ 3) within 4 weeks prior to the first dose.
19. Known human immunodeficiency virus (HIV) infection.
20. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
21. Diagnosed with the other malignancies that may change the expected survival or affect the response evaluation.
22. Unresolved toxicity of previous anti-tumor therapy.
23. History of severe hypersensitivity to inactive ingredients in the drug substance and drug product or other monoclonal antibodies.
24. Have any diseases, medical conditions, organ system dysfunction, or social conditions that may interfere with the subject ability to sign the ICF, adversely affect the subject ability to cooperate and participate in the study, or affect the interpretation of study results, including but not limited to mental illness or substance/alcohol abuse, in the opinion of the investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) by RECIST1.1 and PCWG3 criteria per investigators' review | Approximately within 36 months
  defined as percentage of participants with confirmed best overall response of confirmed complete response (CR) or partial response (PR) to treatment
Radiographic progression free survival (rPFS), and rPFS rate at 3/6 months by RECIST1.1 and PCWG3 criteria per investigators' review | Approximately within 36 months
  defined as the time from the date of first administration to first documented progressive disease (PD) per RECIST1.1 and PCWG3 or death from any cause, whichever occurs first.
Recommended dose of YL201 for the pivotal clinical trial. | Approximately within 36 months

SECONDARY OUTCOMES:
disease control Rate (DCR) by RECIST1.1 and PCWG3 criteria per investigators' review | Approximately within 36 months
  Disease control rate
To evaluate DoR by RECIST1.1 and PCWG3 criteria per investigators' review of YL201 in the treatment of mCRPC | Approximately within 36 months
  Duration of rasponse
To evaluate TTR of YL201 in the treatment of mCRPC | Approximately within 36 months
  Time to Objective response
To evaluate DpR of YL201 in the treatment of mCRPC | Approximately within 36 months
  deepness of response
To evaluate PSA50 response rate and PSA50 response rate at 12 weeks of YL201 in the treatment of mCRPC | Approximately within 36 months
  PSA50 response is defined as a ≥ 50% decline in PSA from baseline with PSA confirmation ≥ 3 weeks after the first documented reduction in PSA of ≥ 50%.
To evaluate TTPR of YL201 in the treatment of mCRPC | Approximately within 36 months
  time to PSA response
To evaluate PDoR of YL201 in the treatment of mCRPC | Approximately within 36 months
  PSA duration of response
To evaluate PDpR of YL201 in the treatment of mCRPC | Approximately within 36 months
  PSA deepness of response
To evaluate TTPP of YL201 in the treatment of mCRPC | Approximately within 36 months
  time to PSA progression
To evaluate TFST of YL201 in the treatment of mCRPC | Approximately within 36 months
  time to first subsequent therapy
To evaluate rPFS of YL201 in the treatment of mCRPC | Approximately within 36 months
  Radiographic Progression Free Survival
To evaluate OS of YL201 in the treatment of mCRPC | Approximately within 36 months
  overall survival
To evaluate time to first symptomatic skeletal event of YL201 in the treatment of mCRPC | Approximately within 36 months
  assessed by investigator according to RECIST v1.1 and PCWG3 criteria
Expression of B7H3 in tumor tissue at baseline and the relationship with the efficacy of YL201. | Approximately within 36 months
Number of participants with AEs, SAEs, and SAEs leading to study treatment interruption or discontinuation. | Approximately within 36 months
  adverse event, serious adverse event
To evaluate the AUC of YL201 | Approximately within 36 months
  the area under curve: AUC is the total amount of YL201 in bloodstream after drug administration
To evaluate the Cmax of YL201 | Approximately within 36 months
  Maximum concentration: The highest measured concentration of YL201 in the bloodstream.
To evaluate the Ctrough of YL201 | Approximately within 36 months
  trough concentration
To evaluate the CL of YL201 | Approximately within 36 months
  Clearance: defined as the amount of drug removed from the bloodstream by the body per unit of time
To evaluate the Vd of YL201 | Approximately within 36 months
  volume of distribution
To evaluate the T1/2 of YL201 | Approximately within 36 months
  Terminal half-life: defined as the time it takes for the concentration of the drug in plasma or serum to be reduced by 50%
To evaluate the E-R relationship of YL201 | Approximately within 36 months
  exposure-response
To evaluate the immunogenicity of YL201 | Approximately within 36 months

CONTACTS AND LOCATIONS:
Locations (24):
- China (24):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Hunan Cancer Hospital, Hunan, Changsha
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital of Huazhong University of Science and Technology Tongji Medical College, Wuhan, Hubei
  - Nanjing Drum Tower hospital, Nanjing, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Shandong Tumor Hospital, Jinan, Shandong
  - Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Ningbo Yinzhou No.2 Hospital, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Fudan University Shanghai Cancer Center, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided